CLINICAL TRIAL: NCT05748340
Title: Comparative Study Between Modified Millard and Mishra Technique in Unilateral Cleft Lip Repair: a Randomised Controlled Study
Brief Title: Unilateral Cleft Lip Repair : Modified Millard and Mishra Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Salah Ahmed, Lecturer pediatric surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-40-2021
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cleft Lip
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): 21normal infant aged 3-6 months
  Interventions: Procedure: Unilateral cleft lip repair
- Group a (Other): 21 patient of unilateral cleft lip had mishra technique repair
  Interventions: Procedure: Unilateral cleft lip repair
- Group b (Other): 21 patient of unilateral cleft lip had modified Millard technique repair
  Interventions: Procedure: Unilateral cleft lip repair

INTERVENTIONS:
Procedure: Unilateral cleft lip repair — Surgical repair unilateral cleft lip

SUMMARY:
Our study findings show that vertical lip length and philtral lip height significantly longer in Millard group than Mishra group in immediate postoperative assessment and nasal width was significantly wider in Mishra group than Millard in 3-month postoperative assessment, This may be attributed to that Mishra group deformity was more severe. The lip shape, the vermilion shape was better in Millard technique than Mishra technique, however, this was statistically insignificant The scar shape was less evident in Mishra technique than Millard technique. But this was also statistically insignificant. However, no major difference in the overall results between the Mishra and Millard rotationadvancement repairs. Thus, either technique could be used for unilateral clefts, as the goal of cleft lip repair is making a symmetrical lip with minimal scar restoring the normal appearance of the face and functional anatomy Anthropometric Measurement of surgical outcome evaluates the surgical technique used and helps to compare between cleft and non-cleft side showing the degree of deformity and we used Subjective assessment to analyse facial aesthetics and appearance impairment as the harmony of a person's face is as Important as measurements, so they should be used together in our opinion.

DETAILED DESCRIPTION:
Cleft lip and palate, which affects 0.5-1.6 out of every 1000 live births, is the most prevalent congenital defect of the head and neck .

When the palatal shelves and the medial nasal process fail to fuse together between the fourth and eighth weeks of development, unilateral cleft lip and palate results . Lip muscles are disrupted and abnormally inserted to the columellar base on the non-cleft side and from the alar base on the cleft side. The nasal floor and alveolus on the cleft side may be deficient or absent. Several approaches, including quadrangular flaps, triangular flaps, and rotationadvancement procedures, were established in the middle of the twentieth century White Roll Vermilion Turn Down Flap (WRV flap) from the lateral lip element Making a symmetrical lip with a small scar and restoring the face's natural appearance and functional structure are the objectives of cleft lip repair . Over the past century, numerous surgical repair approaches have been developed The first known cleft-lip repair was a straight-line suture and a simple cut along the cleft borders, followed by a curved incision to lengthen the lip Drawbacks of straight-line restorations included vertical scar contracture and lip notching Tennison-triangular Randall's approach, which relies on mathematical calculations and lessens vertical lip contraction, is the most popular triangular technique, however the scar violates the philtrum.The Millard rotation-advancement approach was created to align the scar with the philtral column naturally occurring. The initial rotation-advancement technique underwent various variations. Vermilion notching and a scar along the philtral line can be noticed in Millard's repair. The Cupid's bow is distorted and the white roll up is pulled up by scar contracture. was employed by Mishra to modify Millard's technique to create the vermilion and white roll on the medial lip segment. If there is medial hypoplastic vermilion or partial medial vermilion loss, the Mishra procedure is also used Anthropometric Evaluation of surgical technique and comparison of cleft and non-cleft sides are two benefits of measuring surgical outcome .Farkas and colleagues, provided normative measurements of the lip and nose. Qualitative Assessment is subjective assessment and can analyze facial aesthetics and appearance impairment using scales, indices, scoring systems, and rankings. Both direct and indirect techniques can be used to perform anthropometric measurements and qualitative assessments. The most accurate anthropometric method is direct anthropometry, which is the gold standard but requires general anesthesia in young kids. Two dimensional (2D) images can be used for indirect anthropometry; however, calibration and image distance standardization are needed for linear measurements.

ELIGIBILITY:
Inclusion Criteria:

* Infants with unilateral isolated cleft lip aged from 2-6 months
* Infants with incomplete and complete unilateral cleft lip(reach floor of the nose)

Exclusion Criteria:

* Infants less than 2 months or more than 6 months
* Bilateral cleft lip patients
* Recurrent repair cleft lip cases
* Facial cleft cases 5-Syndromic patients cases

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Surgical repair unilateral cleft lip measurements | At 3 months post operative
  1. Vertical lip height
  2. Horizontal lip length
  3. Philtral length

CONTACTS AND LOCATIONS:
Overall Officials: Kasr Elainy, Principal Investigator — Cairo university Egypt
Locations (1):
- Faculty of medicine Cairo university, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Shared for every one
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once publication
Access Criteria: Open for every one